CLINICAL TRIAL: NCT04166188
Title: Lumbar Erector Spinae Plane Block: Cadaveric Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16607219.4.0000.0065
Record Dates: First submitted 2019-11-11; First posted 2019-11-18 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-10

CONDITIONS: Pain; Regional Anesthesia Morbidity; Arthroplasty Complications
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadavers (Experimental): 20ml of 0.01% methylene blue solution (50mg of methylene blue diluted in 0.9% saline 500ml) will be injected, simulating the LESP block technique: injection between the transverse process of the fourth lumbar vertebra (L4) and the erector muscle of the underlying spine.
  The injection will be performed with a Quincke 20G 100-150mm ultrasound-guided needle with a low-frequency curvilinear transducer (4-8 MHz - SonoSite) in the plane between the transverse process of L4 and the spinal erector muscle, bilaterally in each cadaver. by the same operator.
  After injection of the solution the cadavers will be submitted to posterior lumbar region dissection by an anatomist and analyzed the dispersion and impregnation of the blue solution. The anatomical structures with the dye dispersion will be photographed and stored.
  Interventions: Procedure: Lumbar erector spinae plane block

INTERVENTIONS:
Procedure: Lumbar erector spinae plane block — Injection of blue solution in the erector spinae plane in L4 ultrasound-guided and posterior dissection of the lumbar region.

SUMMARY:
Erector spinae plane block (ESP block) was first described by Forero et al for the treatment of neuropathic chest pain. Total hip arthroplasty is a surgery with a high potential for severe postoperative pain, and greater attention should be paid to postoperative analgesia. There are multiple forms of postoperative analgesia for total hip arthroplasty, such as subarachnoid morphine, femoral nerve block, obturator and lateral femoral cutaneous block, lumbar plexus block, continuous epidural block, and "3 in 1" block, for example. ESP (LESP) block has emerged based on the same principle as the ESP block in the thoracic region. So far, to the best of our knowledge, there are only a few case reports that evidence its use for hip surgery analgesia. This study aimed to study the local anesthetic dispersion and the mechanism of action of the blockade.

An experimental, analytical and prospective study will be carried out in which eight fresh adult human cadavers will be selected and injected with 20 ml of 0.01% methylene blue solution at L4 level. The injection will be performed with a Quincke 20G 100-150mm ultrasound-guided needle with a low-frequency curvilinear transducer (4-8 MHz - SonoSite) in the plane between the transverse process of L4 and the spinal erector muscle, bilaterally in each cadaver. by the same operator. After injection of the solution, the cadavers will be submitted to posterior lumbar region dissection by an anatomist and analyzed the dispersion and impregnation of the blue solution.

DETAILED DESCRIPTION:
1. INTRODUCTION

   Erector spinae plane block (ESP block) was first described by Forero et al for the treatment of neuropathic chest pain, in which anesthetic is injected between the spinal erector muscle and the transverse vertebral process in the thoracic region, and in theory, it tends to spread to the anterior paravertebral space, to some vertebral spaces above and below the injection site. However, its mechanism of action and exact local anesthetic dispersion have not yet been fully explained clearly.

   Such blockade, first described for neuropathic chest pain and later expanded for thoracic and abdominal surgery, has shown other applicability, such as cardiac and breast surgeries.

   Forero et al published in July 2018 a study to anatomically demonstrate, from cadaver dissection, the dispersion of dye injected into the same ESP block target at different thoracic levels. They showed the dispersion of methylene blue to the anterior paravertebral space at the injection level in all cadavers, with variable cerebrospinal flow dispersion. In addition there was lateral and medial dispersion to the puncture site, for intercostal spaces, paravertebral sympathetic chain and parietal pleura. However, there are no studies regarding lumbar erector spinae plane block (LESP block) block.

   Since 1960 total hip arthroplasty has become one of the most frequent surgeries in the world, due to its technical revolution with improved quality of life of patients with osteoarthritis, rheumatoid arthritis and proximal femur fractures, for example. However, it is a surgery with high postoperative pain potential, and more attention should be paid to postoperative analgesia, since patients undergoing this type of surgery are usually older patients with multiple comorbidities, more sensitive to adverse effects of systemic analgesic drugs (anti-inflammatory drugs, opioids). In addition, pain may lead to hypomobility, which increases the risk of thromboembolic complications.

   There are multiple forms of postoperative analgesia for total hip arthroplasty, such as subarachnoid morphine, femoral, obturator and lateral femoral cutaneous nerve block, lumbar plexus block, continuous epidural block, and "3 in 1" block, for example. still considered as the gold standard analgesia for such surgery, intrathecal morphine has some adverse effects as burden: pruritus, urinary retention, nausea and vomiting.The "3 in 1" block has a considerable incidence of partial failure, despite being an unique injection block. Blockade of the lateral femoral obturator, obturator, and nerve nerves requires 3 injections and a larger volume of local anesthetic.The epidural technique has the advantage of allowing the use of a long-term epidural catheter, with or without an analgesia-controlled device. (PCA), but in these more fragile patients with multiple comorbidities it may lead to hypotension or limited ambulation due to concomitant use of anticoagulant medications. Lumbar plexus block is a deep block, with greater risk of complications (retroperitoneal hematoma, deep bleeding), of greater technical difficulty, and erratic local anesthetic dispersion.

   The LESP block emerged, based on the same principle as the ESP block in the thoracic region. So far, to the best of our knowledge, there are only a few case reports that evidence its use for hip surgery analgesia. It has potential advantages: ease of execution, low risk of nerve damage and safety in patients with coagulopathies or on anticoagulants. In our service, the investigators have 01 case report presented as a free theme in congress that also describes a good individual effectiveness .

   Recent reports have demonstrated lumbar-level ESP block (LESP) for hip and proximal femur surgery, showing good results in postoperative pain control. One of the first works on lumbar ESP block was a letter to the editor in Tulgar et al's Journal of Clinical Anesthesia, which then began a trial comparing LESP with lumbar square, a work still in progress.

   With the growing interest of anesthesiologists in ESP block, several studies and case reports have been written in different blockade applications, but the literature lacks cadaveric studies to demonstrate more clearly the local anesthetic dispersion and anatomically justify its clinical effectiveness. .
2. BACKGROUND Hip and proximal femur surgeries usually present with significant postoperative pain, which may hinder patient movement and physiotherapy in the postoperative period, besides immobility predisposing to the development of deep vein thrombosis.

   There are several ways of postoperative analgesia for this type of surgery, each having its benefits and harms in relation to the other. This project aims to study the local anesthetic dispersion in the blockade of the lumbar spine erector plane, in order to apply it more safely and effectively as a new modality of analgesia for the hip and proximal femur.
3. OBJECTIVES 3.1. Primary objective The aim of this cadaveric study is to demonstrate the dispersion of methylene blue dye solution when injected into the same anatomical space targeted by the LESP block by anatomical dissection of the lumbar region of cadavers.
4. HYPOTHESIS Lumbar erector spinae plane block (LESP) may provide effective postoperative analgesia for hip and proximal femur surgery, comparable to other existing analgesic modalities. A possible explanation for this is the local anesthetic dispersion injected by this technique, which possibly reaches the posterior lumbar plexus branches.
5. METHODS 5.1 Type of study and scenario An experimental, analytical and prospective study will be conducted at the Capital Death Verification Service (SVOC) and at the Human Anatomy Discipline Laboratory of the University of São Paulo School of Medicine. After approval by the Research Ethics Committee of the School of Medicine of the University of São Paulo, the inclusion of subjects for the study will be initiated.

5.2 Inclusion and exclusion criteria Fresh cadavers, age> 18 years, height between 150cm and 190cm, any gender will be included.

Corpses with severe spinal deformity, known history of lumbar spine surgery, scars suggestive of large anatomical manipulations of the lumbar region, and corpses with BMI> 35 kg / m² will be excluded.

5.3 Sample Calculation Eight cadavers will be used, with injections of solutions simulating the LESP block, bilaterally, totaling 16 injections and dissections.

5.4 Experimental Design 20ml of 0.01% methylene blue solution (50mg of methylene blue diluted in 0.9% saline 500ml) will be injected, simulating the LESP block technique: injection between the transverse process of the fourth lumbar vertebra (L4) and the erector muscle of the underlying spine.

The injection will be performed with a Quincke 20G 100-150mm ultrasound-guided needle with a low-frequency curvilinear transducer (4-8 MHz - SonoSite) in the plane between the transverse process of L4 and the spinal erector muscle, bilaterally in each cadaver. by the same operator.

After injection of the solution the cadavers will be submitted to posterior lumbar region dissection by an anatomist and analyzed the dispersion and impregnation of the blue solution. The anatomical structures with the dye dispersion will be photographed and stored.

ELIGIBILITY:
Inclusion Criteria:

* Fresh cadavers;
* Age> 18 years;
* Height between 150cm and 190cm;
* Any gender.

Exclusion Criteria:

* Corpses with severe spinal deformity;
* Known history of lumbar spine surgery;
* Scars suggestive of large anatomical manipulations of the lumbar region;
* Corpses with BMI> 35 kg / m².

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Blue solution dispersion to the lumbar plexus in cadaver | 7 months
  It will be injected 20ml of blue solution in the lumbar erector spinae plane of adult fresh cadavers, ultrasound guided, with posterior dissection of the lumbar region by a neurosurgeon and the investigators to evaluate the dispersion of the solution to the nerve roots of lumbar plexus, simulating a new anesthetic technique.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim Vieira, Study Director — Faculdade de Medicina da Universidade de São Paulo
Locations (1):
- Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Vidal E, Gimenez H, Forero M, Fajardo M. Erector spinae plane block: A cadaver study to determine its mechanism of action. Rev Esp Anestesiol Reanim (Engl Ed). 2018 Nov;65(9):514-519. doi: 10.1016/j.redar.2018.07.004. Epub 2018 Aug 27. English, Spanish. PMID 30166123
- [Result] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Result] Adhikary SD, Pruett A, Forero M, Thiruvenkatarajan V. Erector spinae plane block as an alternative to epidural analgesia for post-operative analgesia following video-assisted thoracoscopic surgery: A case study and a literature review on the spread of local anaesthetic in the erector spinae plane. Indian J Anaesth. 2018 Jan;62(1):75-78. doi: 10.4103/ija.IJA_693_17. PMID 29416155
- [Result] Hamilton DL, Manickam B. The Erector Spinae Plane Block. Reg Anesth Pain Med. 2017 Mar/Apr;42(2):276. doi: 10.1097/AAP.0000000000000565. No abstract available. PMID 28207652
- [Result] Foss NB, Kristensen MT, Palm H, Kehlet H. Postoperative pain after hip fracture is procedure specific. Br J Anaesth. 2009 Jan;102(1):111-6. doi: 10.1093/bja/aen345. PMID 19059921
- [Result] Ibrahim MS, Twaij H, Giebaly DE, Nizam I, Haddad FS. Enhanced recovery in total hip replacement: a clinical review. Bone Joint J. 2013 Dec;95-B(12):1587-94. doi: 10.1302/0301-620X.95B12.31303. PMID 24293586
- [Result] Liang C, Wei J, Cai X, Lin W, Fan Y, Yang F. Efficacy and Safety of 3 Different Anesthesia Techniques Used in Total Hip Arthroplasty. Med Sci Monit. 2017 Aug 2;23:3752-3759. doi: 10.12659/msm.902768. PMID 28767640
- [Result] Kearns RJ, Macfarlane AJ, Anderson KJ, Kinsella J. Intrathecal opioid versus ultrasound guided fascia iliaca plane block for analgesia after primary hip arthroplasty: study protocol for a randomised, blinded, noninferiority controlled trial. Trials. 2011 Feb 21;12:51. doi: 10.1186/1745-6215-12-51. PMID 21338492
- [Result] Kang H, Ha YC, Kim JY, Woo YC, Lee JS, Jang EC. Effectiveness of multimodal pain management after bipolar hemiarthroplasty for hip fracture: a randomized, controlled study. J Bone Joint Surg Am. 2013 Feb 20;95(4):291-6. doi: 10.2106/JBJS.K.01708. PMID 23302898
- [Result] Tulgar S, Senturk O. Ultrasound guided Erector Spinae Plane block at L-4 transverse process level provides effective postoperative analgesia for total hip arthroplasty. J Clin Anesth. 2018 Feb;44:68. doi: 10.1016/j.jclinane.2017.11.006. Epub 2017 Nov 14. No abstract available. PMID 29149734